CLINICAL TRIAL: NCT03534063
Title: Implementing Genomics in Practice (IGNITE): CYP2D6 Genotype-Guided Pain Management in Patients Undergoing Arthroplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of Florida Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201800445; UL1TR001427-04 (NIH); OCR17562 (Other: Universiy of Florida)
Record Dates: First submitted 2018-05-10; First posted 2018-05-23 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Pain, Postoperative
Keywords: Arthroplasty Surgery; Genotype-Guided Pain Management
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CYP2D6-guided opioid therapy (Active Comparator): Participants randomized to the CYP2D6-guided arm will have their CYP2D6 genotyping completed prior to surgery (in the absence of any genotyping error) with results reported in the electronic health record (EHR). Patients will be categorized as CYP2D6 PM, IM, NM, or UM based on CYP2D6 genotype/activity score and FDA guidance on drug interactions. Strong inhibitors (e.g. bupropion, fluoxetine, paroxetine) phenoconvert patients to PMs, with moderate inhibitors (e.g. duloxetine, fluvoxamine) reducing CYP2D6 activity scores by 50%.
  Interventions: Genetic: CYP2D6-guided opioid therapy
- Usual Care (No Intervention): Participants randomized to the usual care arm will have their DNA collected at the start of the study and stored at the lab until after they have completed their surgery and the 2-week follow-up, at which time, their sample was genotyped with the results reported in the EHR.

INTERVENTIONS:
Genetic: CYP2D6-guided opioid therapy — Using a standardized consult note, recommendations were made to avoid tramadol, hydrocodone, codeine, and oxycodone in PMs, IMs, and UMs and to use an alternative opioid (e.g. morphine, hydromorphone) or non-opioid (e.g. NSAID). Consideration of tramadol as the first-line opioid will be recommended for NMs.
  Arms: CYP2D6-guided opioid therapy

SUMMARY:
This will be a randomized, open-labeled pilot pragmatic clinical trial. Patients undergoing arthroplasty surgery will be recruited from the University of Florida (UF) Health Gainesville and the Villages Orthopedic clinics for CYP2D6 pharmacogenetic testing to manage post-surgical pain. Patients will be randomized 2:1 to either usual care or genotype-guided care. The aims of the study were to: 1) test the feasibility of a genotype-guided opioid prescribing approach for patients undergoing an outpatient surgical procedure, a group at high risk for persistent opioid use; and 2) evaluate the effect of genotype-guided post-surgical pain management on pain control and opioid prescribing.

DETAILED DESCRIPTION:
This study was a randomized, open-label, type 2 hybrid implementation effectiveness trial conducted to test the hypothesis that CYP2D6 genotype-guided management of post-surgical pain 1) was feasible, and 2) reduced the use of codeine, tramadol, hydrocodone, and oxycodone in Poor Metabolizers (PMs), Intermediate Metabolizers (IMs), and Ultrarapid metabolizers (UMs). In addition to the reduced use of opioids listed above, we aimed to see if participants had improved post-operative pain control in PMs/IMs and reduced Drug Enforcement Administration (DEA) Schedule II (C-II) opioids in Normal Metabolizers (NMs). Patients scheduled to undergo arthroplasty surgery were recruited from the UF Health Gainesville and the Villages Orthopedic clinics. Patients were randomized 2:1 to a genotype-guided versus usual care approach. For patients with CYP2D6 PM, IM or UM phenotype based on genotype or drug interactions, a recommendation to avoid hydrocodone, tramadol, codeine, and oxycodone were made. In NMs, tramadol was recommended, given evidence of its lower potential addiction risk than C-II opioids. Patient-Reported Outcomes Measurement Information System (PROMIS) measures were administered at baseline (within 30 days of surgery) and 2 weeks ± 4 days post-surgery for patients in each arm. Pain scores and assessments of physical functioning, emotional functioning, and mobility from the PROMIS measures and utilization of pain medications during the 2-week period following surgery were also compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo total joint arthroplasty at area hospital
* Primary unilateral total hip or knee arthroplasty scheduled within approximately 6 months of the initial evaluation clinic visit

Exclusion Criteria:

* Patients scheduled to undergo a revision or bilateral procedure
* Receiving chronic opioid therapy, defined as the use of opioids on most days for > 3 month
* Allergy to opioids

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larisa Cavallari, PharmD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - UF Health at the University of Florida, Gainesville, Florida
  - Unversity of Florida, Gainesville, Florida
  - UF Health Orthopaedic--Villages, Summerfield, Florida

REFERENCES:
- [Result] Thomas CD, Parvataneni HK, Gray CF, Deen JT, Prieto HA, Pulido LF, Elsey AR, Elwood EN, Starostik P, Gong Y, Fillingim RB, Johnson JA, Cavallari LH. A hybrid implementation-effectiveness randomized trial of CYP2D6-guided postoperative pain management. Genet Med. 2021 Apr;23(4):621-628. doi: 10.1038/s41436-020-01050-4. Epub 2021 Jan 8. PMID 33420349

RESULTS

PARTICIPANT FLOW:
Groups:
- Genotype-guided Opioid Therapy: For participants randomized to the genotype-guided arm, a CYP2D6 phenotype and pharmacist consult note will be provided to physicians to assist in opioid prescribing.
- Usual Care: For participants randomized to the usual care arm, providers will follow usual care prescribing practices for post operative opioid prescribing.
Period: Overall Study
Arm/Group | Genotype-guided Opioid Therapy | Usual Care
Started | 173 | 87
Completed | 154 | 80
Not Completed | 19 | 7

BASELINE CHARACTERISTICS:
Population: Overall number of baseline participants analyzed were participants who were enrolled, randomized, and completed arthroplasty joint surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | Genotype-guided Opioid Therapy | Usual Care | Total
Number analyzed (Participants) | 154 | 80 | 234
Age, Categorical [Count of Participants; unit: Participants] — Population: The participants included in the analysis were the ones who received the allocated intervention (surgery).
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 61 | 40 | 101
    >=65 years | 93 | 40 | 133
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The participants included in the analysis were the ones who received the allocated intervention (surgery).
  Participants
    Female | 91 | 46 | 137
    Male | 63 | 34 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The participants included in the analysis were the ones who received the allocated intervention (surgery).
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 3 | 1 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 16 | 12 | 28
    White | 131 | 65 | 196
    More than one race | 4 | 2 | 6
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: The participants included in the analysis were the ones who received the allocated intervention (surgery).
  Participants
    United States | 154 | 80 | 234

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Agreed to Participate
Description: The feasibility of clinical implementation was measured by the percentage of approached patients who agreed to be the study. This was measured by the number of patients approached and the number of patients who enrolled in the study.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Participants Approached for the Study, Prior to Randomization: Total count of participants approached to enroll into the study, prior to randomization.
Arm/Group | Participants Approached for the Study, Prior to Randomization
Number analyzed (Participants) | 282
Participants
  Agreed to participant and enrolled into the study | 260
  Declined to participant in the study | 22

2. Primary Outcome: Percentage of Participants With a Clinical Phenotype Warranting Alternative Therapy
Description: The feasibility of implementing a genotype-guided opioid prescribing approach for participants undergoing an elective surgical procedure was analyzed by the percentage of participants in the genotype-guided arm and usual care arm with a high-risk CYP2D6 phenotype. CYP2D6 phenotypes were based on CYP2D6 genotype and phenoconversion. High-risk CYP2D6 phenotypes were poor metabolizers (PM), intermediate metabolizers (IM), ultrarapid metabolizers (UM), and ranged phenotypes such as normal to ultrarapid metabolizers and intermediate to ultrarapid metabolizers.
Time Frame: An average of 2 weeks after genotype sample collection
Population: Participants enrolled and randomized who underwent a total joint arthroplasty procedure, completed the study, and were genotyped.
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype-guided Opioid Therapy | Usual Care
Number analyzed (Participants) | 154 | 74
Participants
  High-Risk CYP2D6 Phentoype | 35 | 28
  Normal CYP2D6 Phenotype | 119 | 46

3. Primary Outcome: Percentage of Participants in the Genotype-guided Arm for Whom a Clinical Phenotype-guided Recommendation Was Accepted by the Clinician
Description: The feasibility of clinical implementation was measured by the percentage of participants in the genotype-guided arm for whom a clinical phenotype-guided recommendation was accepted by the clinician. Study recommendations were considered accepted for participants with a high-risk phenotype if an alternative opioid (e.g., hydromorphone, morphine) was prescribed. For CYP2D6 normal metabolizers (NM), consult recommendations were accepted if tramadol was prescribed. Participants were typically prescribed a tramadol-based regimen where in most cases hydrocodone, or another opioid, was prescribed concomitantly with tramadol as is usual practice at the clinics where participants were enrolled. Participants whose genotype resulted after the preoperative appointment were excluded from the analysis of acceptance of consult recommendations. Data for this outcome were only collected from participants in the genotyped-guided arm with CYP2D6 results returned prior to the preoperative appointment.
Time Frame: An average of 2 months after genotype results returned
Population: Participants in the genotyped-guided arm with CYP2D6 results returned prior to the preoperative appointment.
Measure: Count of Participants; unit: Participants
Groups:
- High-Risk CYP2D6 Phenotype in the Genotype-guided Arm: Participants in the Genotype-guided arm and those with genotype returned prior to the preoperative appointment that had a high-risk (IM/PM/UM/NM-UM) CYP2D6 phenotype.
- Normal CYP2D6 Phenotype in the Genotype-guided Arm: Participants in the genotype-guided arm and those with genotype returned prior to the preoperative appointment that had a normal CYP2D6 phenotype.
Arm/Group | High-Risk CYP2D6 Phenotype in the Genotype-guided Arm | Normal CYP2D6 Phenotype in the Genotype-guided Arm
Number analyzed (Participants) | 29 | 115
Participants | 21 | 101

4. Primary Outcome: Opioid Utilization
Description: Opioid consumption was calculated as the difference between participant-reported opioid pills prescribed at the preoperative appointment and opioid pills remaining at the 2-week time point. This difference was calculated for each opioid and then expressed as morphine milligram equivalents (MME) using standard conversion factors and the medication strength of the prescribed opioid analgesic. If a participant was prescribed multiple opioids, MMEs were calculated for each opioid and then summed to give a total MME value.
Time Frame: 2 weeks after surgery
Population: Study population that completed a 2-week post-surgery follow-up survey.
Measure: Mean (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Genotype-guided Opioid Therapy | Usual Care
Number analyzed (Participants) | 126 | 68
morphine milligram equivalents | 200 [104 to 280] | 230 [133 to 350]
Statistical Analysis 1: Comparison: Genotype-guided Opioid Therapy vs Usual Care; Test type: Superiority; p = .047, Wilcoxon (Mann-Whitney); Comparisons for opioid consumption and composite pain intensity were performed by analysis of covariance, adjusting for baseline differences in groups

5. Secondary Outcome: Composite Pain Intensity
Description: Composite pain intensity was compared between the genotype-guided arm and usual care arm 2 weeks after surgery. The first two scales in the PROMIS Pain Intensity item bank assess pain intensity utilizing a 7-day recall period (items include the phrase "the past 7 days") while the third scale asks the patient to rate their pain intensity "right now." Each of the 3 scales (worst pain, average pain, and current pain) used to calculate the composite pain intensity score has a range of 1 to 5, with the following text assigned to the numeric scale, 1 -"had no pain", 2 -"mild", 3 -"moderate", 4 -"severe", and 5 -"very severe." The mean composite pain intensity ranges from 1-5. The higher the composite pain score, the more pain and thus worse outcomes.
Time Frame: 2 weeks after surgery
Population: Participants that completed the pain intensity survey 2 weeks after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CYP2D6-guided Opioid Therapy | Usual Care
Number analyzed (Participants) | 137 | 74
units on a scale | 2.6 (0.8) | 2.5 (0.7)
Statistical Analysis 1: Comparison: CYP2D6-guided Opioid Therapy vs Usual Care; Test type: Superiority; p = .638, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected as a part of this study.
Description: Opioid-related adverse events were not systematically collected as part of the study.
Groups:
- Genotype-guided Opioid Therapy: The study team will collect data on the implementation success metrics, patient-reported outcomes with Patient-Reported Outcomes Measurement Information System (PROMIS) measures, and opioid utilization measures. The investigators will collect a proportion of patients prescribed specific opioids and self-reported opioid use, since patients may not take any or all of the opioids prescribed.
  CYP2D6-guided post-operative: For patients randomized to the genotype-guided arm, saliva or buccal cell sample will be collected unless venipuncture is done for other reasons and then a blood sample will be collected for genotyping.
- Usual Care: The study team will collect data on the implementation success metrics, patient-reported outcomes with Patient-Reported Outcomes Measurement Information System (PROMIS) measures, and opioid utilization measures. The investigators will collect a proportion of patients prescribed specific opioids and self-reported opioid use, since patients may not take any or all of the opioids prescribed.
Arm/Group | Genotype-guided Opioid Therapy | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Assessment of MME may be considered exploratory. Reliance on participant reported opioid consumption restricts MME analysis to those who successfully completed the two-week survey. Participants could have received any number of analgesics at various doses, reliance on participant responses was key to calculating MME at the follow-up timepoints, and incomplete participant-reported data reduces the available sample to assess postoperative opioid consumption.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT03534063/Prot_SAP_ICF_000.pdf